CLINICAL TRIAL: NCT02809625
Title: Application of Dynamic Contrast Enhanced MRI in Clinical and Early Diagnosis of Brucellar Spondylitis
Brief Title: Application of DCE-MRI in the Diagnosis of Brucellar Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Inner Mongolia Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: AHInnerMongolia
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Brucella Spondylitis
Keywords: Dynamic contrast -enhanced MRI; brucella spondylitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Brucellosis, also known as Mediterranean fever, undulant fever, or Malta fever is a zoonotic disease caused by Brucella infection.With the rapid development of animal husbandry and aquaculture and increasing consumption of dairy products in urban residents, the incidence of this disease in Inner Mongolia and even in the mainland area of China is significantly increased.

The disease can damage multiple systems including nervous system, circulatory system, reproductive system and bone joints, etc. The sooner the diagnosis of brucellar spondylitis is diagnosed and treated, the better will be the prognosis of the patients which can prevent the development of severe complications and diminish the need for surgical therapy. Thus the early diagnosis of brucellar spondylitis was of great significance.We quantitatively analyzed the brucellar spondylitis with DCE-MRI to explore the application of DCE-MRI in the early diagnosis of brucellar spondylitis.

DETAILED DESCRIPTION:
About 100 patients with Brucellosis were conducted with conventional MRI and dynamic contrast-enhanced MRI(DCE-MRI) scan. The variations of the value of ktrans（endothelial transfer constant），kep（reflux rate）,Ve(fractional extracellular fluid space volume) and Vp(fractional plasma volume) between the vertebral lesions,Early lesions of vertebral body and normal tissues were measured and compared. And under the receiver operating characteristic（ROC） curve analysis,we will calculate the sensitivity and specificity of Ktrans,Kep,Ve and Vp in the diagnosis and early diagnosis of brucella spondylitis .The values of Ktrans,Kep,Ve and Vp will be studied between the vertebral lesions and normal tissues, the early lesions of vertebral body and normal tissues.The sensitivity and specificity of both parameters (Ktrans、Kep、Ve、Vp)will be done.The valve of DCE-MRI in the diagnosis and early diagnosis of the brucella spondylitis will be analysed.

ELIGIBILITY:
Inclusion Criteria:

The epidemiological exposure history of different extents, accompanied with symptoms including

* low fever
* night sweats
* intermittent lower back pain
* movement limitation

Exclusion Criteria:

* With other disease like tuberculous spondylitis,vertebral metastases,etc

Ages: 35 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: About 100 patients with Brucellosis including patients with brucella spondylitis obviously and patients with obvious waist pain but the conventional MRI showed no obvious abnormalities were selected.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The useful value of dynamic contrast-enhanced MRI in clinical diagnosis and early diagnosis of brucella spondylitis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peng fei Qiao, MD, Study Director — The Affiliated Hospital of Inner Mongolia Medical University
Locations (1):
- The Affiliated Hospital of Inner Mongolia Medical University, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided